CLINICAL TRIAL: NCT02705417
Title: Maximizing Native Arteriovenous Fistulae Rates. Is Routine Colour Doppler Vascular Mapping in Pre-operative Planning of Value? A Retrospective Study.
Brief Title: Maximizing Native Arteriovenous Fistulae Rates.
Status: Completed | Type: Observational
Sponsor: Medifil AE (Other)
Collaborators: International Renal Research Institute Vicenza (Other)
Responsible Party: Principal Investigator, Ioannis Emmanouel Giannikouris, Assistant for the Medical Director, Medifil AE
Other Study IDs: 1
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Failure; Arteriovenous Shunt; Hemodialysis
Keywords: arteriovenous fistula; colour Doppler; physical examination; renal dialysis; retrospective studies
MeSH Terms: conditions — Renal Insufficiency; Arteriovenous Fistula | interventions — Restraint, Physical; Health Records, Personal; Polytetrafluoroethylene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients in whom selection of vascular access relied upon physical examination and medical history, during pre-operative surgical assessment
  Interventions: Procedure: physical examination; Procedure: medical history; Procedure: native arteriovenous fistula construction; Procedure: arteriovenous graft placement
- Group B: Patients who underwent vascular mapping using color Doppler Ultrasonography in addition to physical examination and history during pre-operative evaluation.
  Interventions: Procedure: preoperative color Doppler ultrasonographic vascular mapping; Procedure: physical examination; Procedure: medical history; Procedure: native arteriovenous fistula construction; Procedure: arteriovenous graft placement

INTERVENTIONS:
Procedure: preoperative color Doppler ultrasonographic vascular mapping — Preoperative color Doppler ultrasonographic vascular mapping was performed with linear probe. The patient extremity under scrutiny was placed under support, with tourniquet augmentation. Vessels were examined in both short (transverse) and long (longitudinal) axis. Anatomical variations, wall morphology and internal diameters at the antecubital fossa, the proximal (cranial), mid and distal (caudal) third of the arm and forearm were assessed in both extremities. Veins were evaluated for compressibility and adequate drainage to deep venous system. The presence of sclerotic, thrombosed and fibrosed segments were noted. Doppler waveforms were obtained in the long axis and volume flow (VF) calculated for arteries selected for potential access construction.
  Other Names: vascular mapping; pre-operative mapping
  Groups: Group B
Procedure: physical examination — Arterial pulse examination, differential blood pressure measurements and the Allen test in both extremities. Inspection of the superficial venous system with tourniquet enhancement in the arm was performed during venous assessment.
  Other Names: clinical examination
Procedure: medical history — medical history with respects to diabetes mellitus, coronary heart disease, peripheral vascular disease
Procedure: native arteriovenous fistula construction — surgigal creation of native arterial and venous anastomoses
Procedure: arteriovenous graft placement — surgical placement of arteriovenous graft
  Other Names: Polytetrafluoroethylene (PTFE) synthetic graft

SUMMARY:
The purpose of our study is to compare physical examination alone to color Doppler ultrasonography (CDUS) vascular mapping and physical examination in terms of outcomes of vascular access and long-term patency.

DETAILED DESCRIPTION:
Fistula maturation is a complex vascular remodelling process that requires vessel dilation, increases in volume flow rates in the feeding artery and afferent vein and structural alterations of the vascular wall. The understanding of these procedures and the factors involved in promoting maturation is limited. In this context, one of the major areas requiring investigation is the identification of clinically useful pre-operative predictors of access outcome.

Traditionally, the selection of vascular access and the eligibility for native arteriovenous fistula construction was mainly determined by findings of clinical examination. However, in addition to a complete history and physical examination, National Kidney Foundation/Dialysis Outcome Quality Initiative (NFK/DOQI) recommended that routine pre-operative color Doppler ultrasonographic vascular mapping should be performed in all hemodialysis patients who are candidates for access formation. This concerns the routine implementation of a non-invasive, safe and cost-effective method that permits the identification of vessels that are suitable for arteriovenous fistula (AVF) construction, acknowledging that supporting Level I evidence is still lacking. Indeed, available data supporting the significance of mapping on access maturation and patency rates are limited and conflicting.

The aim of the present study is to compare the type of preoperative assessment, physical examination alone to combined CDUS vascular mapping and physical examination, to outcomes of performed vascular access procedures with respect to type selection and long-term patency at 12 months in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease

Exclusion Criteria:

* poor life expectancy
* congestive heart failure New York Heart Association stage 3 and over
* candidates for tunneled catheters

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dialysis dependent end stage renal disease with first time permanent vascular access, more specifically native arteriovenous fistula or arteriovenous grafts.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
number of native AVF constructed | in 1 month

SECONDARY OUTCOMES:
primary patency rates | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis E. Giannikouris, PhD, Principal Investigator — Medifil AE Private Hemodialysis Centre

IPD SHARING:
Plan to Share IPD: Yes